CLINICAL TRIAL: NCT04289818
Title: Efektivitas "CARE Coaching Model" Sebagai Upaya Pemberdayaan Pasien Diabetes Untuk Meningkatkan Status Kesehatan Dan Perilaku Pengendalian Diabetes
Brief Title: The Effectiveness of "CARE Coaching Model" as an Effort to Empower Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Prof. Dr. dr. Pradana Soewondo, SpPD-KEMD, Professor, Endocrinologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PS002
Record Dates: First submitted 2020-02-10; First posted 2020-02-28 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Type 2
Keywords: Diabetes Mellitus; Health coaching
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Conventional Education Class
- Coaching (Experimental): Health Coaching
  Interventions: Other: Health Coaching

INTERVENTIONS:
Other: Health Coaching — Health Coaching as face to face with a coach
  Arms: Coaching

SUMMARY:
In Indonesia and others countries, only 30.8% patients with type 2 diabetes mellitus (T2DM) achieved glycemic control with HbA1c <7%. Optimal pharmacological treatment alone does not guarantee an optimal outcome, therefore it should be combined with lifestyle management. Health coaching helps T2DM patients increase self awareness to improve and maintain behavior which play a role in self-management. This study aims to evaluate the impact of health coaching on glycemic control on T2DM patients.

DETAILED DESCRIPTION:
Subjects randomized into 2 groups: control and intervention group. All subject received education class in top of standard treatment. Intervention group received additional personal health coaching.

Education and health coaching was given for 12 sessions every 2 weeks with 12 different themes for each session. Health coaching were given by International certified health coach.

Laboratory examination and questionnaire collected at baseline, 3 and 6 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* T2DM patients
* aged 30-60 years old
* HbA1C > 7.5% within the past 3 months
* able to write and read.

Exclusion Criteria:

* Patients with cognitive disease (such as dementia)
* having hearing problem or sight problem
* unable to live independently on daily basis
* having disease that may affect HbA1c result (eg: hemolytic anemia)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline HbA1c at 3 months | 3 month after intervention
  Glycemic Control
Change from Baseline HbA1c at 6 months | 6 month after intervention
  Glycemic Control

SECONDARY OUTCOMES:
Change from Baseline Fasting Plasma Glucose at 3 months | 3 month after intervention
  Glycemic Control
Change from Baseline 2-hours post prandial plasma glucose at 3 months | 3 months after intervention
  Glycemic control
Change from HDL-cholesterol at 3 months | 3 months after intervention
  Diabetes mellitus control
Change from LDL-cholesterol at 3 months | 3 months after intervention
  Diabetes mellitus control
Change from Triglycerides at 3 months | 3 months after intervention
  diabetes mellitus control
Change from Total Cholesterol at 3 months | 3 months after intervention
  Diabetes mellitus control
Change of Body mass index at 3 months | 3 month after intervention
  Diabetes mellitus control
Change calorie intake at 3 months | 3 month after intervention
  life style parameter
International Physical Activity Questionnaire (IPAQ) questionnaire | baseline, 3 month and 6 months after intervention
  consist of several question about activities in the whole week. Scoring divided into 3 categories : low, moderate, high. This questionnaire is to describe activities no to divided whether high score means good or bad
EQ-5D quality of life questionnaire | baseline, 3 month and 6 months after intervention
  This questionnaire consist of several question with 5 main outcome mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Subjects will answer the question with fully, half or none.
Change from Baseline Fasting Plasma Glucose at 6 months | 6 month after intervention
  Glycemic Control
Change from Baseline 2-hours post prandial plasma glucose at 6 months | 6 months after intervention
  Glycemic Control
Change from HDL-cholesterol at 6 months | 6 months after intervention
  diabetes mellitus Control
Change from LDL-cholesterol at 6 months | 6 months after intervention
  diabetes mellitus Control
Change from Triglycerides at 6 months | 6 months after intervention
  diabetes mellitus Control
Change from Total Cholesterol at 6 months | 6 months after intervention
  diabetes mellitus Control
Change from systolic and diastolic blood pressure at 6 months | 6 months after intervention
  diabetes mellitus Control
Change calorie intake at 6 months | 6 months after intervention
  life style parameter
Change of Body mass index at 6 months | 6 months after intervention
  diabetes mellitus control

CONTACTS AND LOCATIONS:
Overall Officials: Pradana Soewondo, Prof, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia